CLINICAL TRIAL: NCT06077383
Title: Effect of Weizmania Coagulans BC99 Intervention on Gut Microbiota and Metabolic Markers in Overweight/Obese Adults: Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Weizmania Coagulans BC99 Intervention on Gut Microbiota and Metabolic Markers in Overweight/Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QLYY-202307-008
Record Dates: First submitted 2023-09-08; First posted 2023-10-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2023-09

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): Probiotics group subjects take probiotics every day for 8 weeks.
  Interventions: Dietary Supplement: Weizmania Coagulans BC99
- Placebo group (Placebo Comparator): Placebo group subjects take placebo every day for 8 weeks.
  Interventions: Dietary Supplement: Weizmania Coagulans BC99

INTERVENTIONS:
Dietary Supplement: Weizmania Coagulans BC99 — Probiotics group subjects take probiotics every day for 8 weeks.
  Other Names: placebo

SUMMARY:
The main purpose of this study is to verify the effects of Weizmania Coagulans BC99 on the gut microbiota and fat related markers (TG, TC, HDL, LDL) in overweight/Obese adult subjects.

The subjects participate were randomly grouped and receive intervention with Weizmann clotting bacteria BC99 or placebo. The total duration of the study is 8 weeks. After the intervention, blood, urine, and feces samples of the subjects need to be collected and promptly tested in the laboratory. During the intervention period, each group of subjects was required to take the corresponding product daily and record complications.

DETAILED DESCRIPTION:
The main purpose of this study is to verify the effects of Weizmania Coagulans BC99 on the gut microbiota and fat related markers (TG, TC, HDL, LDL) in overweight/Obese adult subjects.

The subjects participate in the screening on a voluntary basis, and those who pass the screening will enter the trial. Randomly group and receive intervention with Weizmann clotting bacteria BC99 or placebo. The total duration of the study is 8 weeks, including 1 week before the trial (followed up once), 4 weeks during the trial (followed up once a week), and 8 weeks during the trial (followed up once a week). After the intervention, blood, urine, and feces samples of the subjects need to be collected and promptly tested in the laboratory. During the intervention period, each group of subjects was required to take the corresponding product daily and record complications.

ELIGIBILITY:
Inclusion Criteria:

1. All patients meet the diagnostic criteria for severe illness, and a body mass index (BMI) of ≥ 24kg/m2 is considered overweight;
2. Age 18-65 years old;
3. Without dieting or weight loss, and able to accept dietary intervention, maintain a low-carbon and healthy diet during the trial period;
4. Patients who understand clinical research and commit to complying with research requirements and procedures;
5. Patients who have signed informed consent forms. Able to complete research according to the requirements of the experimental protocol;

Exclusion Criteria:

1. Taking items with similar functions to the test subjects in the short term can affect the judgment of the results;
2. Have taken antibiotics 2 weeks before recruitment;
3. Those who stop taking the test sample or add other drugs midway, and cannot determine the efficacy or have incomplete information;
4. Obesity caused by drug treatment (hormones, antidepressants, etc.), endocrine diseases, combined with severe liver and kidney dysfunction, water retention or muscle development;
5. Patients who are pregnant, lactating, stomatal, critically ill, or have potential health conditions that affect metabolism or weight;
6. Neuroendocrine system diseases (hypothyroidism, polycystic ovary syndrome, Cushing's syndrome, hypothalamic injury, etc.);
7. Have a clear history of gastrointestinal diseases (such as ulcers, gastrointestinal bleeding, irritable bowel syndrome, celiac disease, inflammatory bowel disease, Crohn's disease, or other diseases) and a history of surgery (such as weight loss surgery, bandaging surgery, gastrointestinal anastomosis surgery, and intestinal resection surgery);
8. Hereditary obesity Hereditary obesity (such as PWS, Down's syndrome), metabolic obesity (such as obesity reproductive impotence syndrome), endocrine obesity (such as Kirschner's syndrome, hypothyroidism), any disease affecting liver fibrosis or steatosis, metabolic disease (such as hypothyroidism/hyperthyroidism, type 1 or type 2 diabetes, etc.);
9. Patients who changed their diet type during the study period;
10. Patients with severe diseases such as cardiovascular, cerebrovascular, liver, kidney, and hematopoietic systems, as well as endocrine diseases, and mental illnesses;
11. According to the researcher's judgment, the condition of the subject does not qualify them to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
The gut microbiota were sequenced by 16s high-throughput sequencing. | 0, 4 and 8 week
  Verification of the effects of Weizmania Coagulans BC99 on the gut microbiota in overweight adult subjects.

SECONDARY OUTCOMES:
The fat related biomarkers (TG, TC, HDL, LDL) were detected by blood biochemistry. | 0, 4 and 8 week
  Verification of the effects of Weizmania Coagulans BC99 on the fat related biomarkers (TG, TC, HDL, LDL) in overweight adult subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang R, Zhang G, Wang X, Xing Z, Li Z, Li L. Effect of Bacillus coagulans BC99 supplementation on body weight and gut microbiota in overweight and obese individual: a randomized, double-blind, placebo-controlled study. Front Nutr. 2025 May 9;12:1542145. doi: 10.3389/fnut.2025.1542145. eCollection 2025. PMID 40416368